CLINICAL TRIAL: NCT00485238
Title: EFFECTS OF IMMEDIATE ARGON LASER PERIPHERAL IRIDOPLASTY Versus CONVENTIONAL SYSTEMIC MEDICAL THERAPY ON OPTIC NERVE HEAD STRUCTURE AND FUNCTION OF ACUTE PRIMARY ANGLE CLOSURE EYES
Brief Title: ALPI vs Medical Therapy Effects on Optic Nerve Structure & Function
Acronym: Iridoplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Paul TK Chew, A/Prof, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSRB A/06/177
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Glaucoma
Keywords: glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Argon laser Iridoplasty
Drug: Intravenous acetazolamide

SUMMARY:
The aim is to determine which approach, immediate argon laser peripheral iridoplasty or conventional systemic medical treatment efficiently breaks acute angle closure attack without consequent visual morbidities. The specific objectives are to see whether sudden intraocular pressure(IOP) lowering brought about by laser iridoplasty or medical treatment affects optic nerve head structure and function and identify if immediate decompression is associated with greater incidence of ocular problems like corneal endothelial compromise, optic disc edema, macular edema, decompression retinopathy, cataract formation, progression to chronic angle closure.

DETAILED DESCRIPTION:
Primary Angle Closure Glaucoma (PACG) continues to be a major concern in Asia. It is a major cause of visual morbidity in the region1 being the most prevalent type of glaucoma especially in Chinese and Mongoloid descent.2,3 During the acute stage of the disease, prompt institution of measures to break the attack is necessary. Two recognized approaches are utilized in practice in lowering intraocular pressure and preparing for the definitive treatment of laser peripheral iridotomy. These are conventional topical and systemic medical therapy and immediate peripheral iridoplasty using either argon or diode lasers.

In the study of Lim, Tan, Chew, Seah et al., laser iridoplasty was noted to have a useful role in the management of medically unresponsive acute angle closure, particularly in those cases where laser peripheral iridotomy (PI) could not be successfully performed4 . Randomized controlled trials of Lam, Lai, Tham et al. comparing immediate laser peripheral iridoplasty plus topical medications and topical and systemic medical treatment found no significant difference in the eventual mean IOP and requirement for glaucoma medications 5 . However, significant difference in efficacy was observed between the two treatment arms within the first two hours of treatment with argon laser peripheral iridoplasty and topical medications lowering IOP faster than conventional medications6. In all the trials cited, there was no mention of sudden IOP lowering effects of either argon laser iridoplasty or conventional medications on the optic nerve head and visual field status, as well as its effect on other ocular structures like the cornea, lens and retina . In our literature search, two papers studied the optic nerve head structure and function in angle closure glaucoma, but not in the immediate period of sudden IOP lowering. Ang, Aung, Chua, Yip and Chew made a comparative assessment of the visual field loss between symptomatic and asymptomatic PACG, with 50% of asymptomatic PACG subjects presenting with end stage visual field loss in contrast to just 7% of symptomatic PACG.7 Lai, Tham, Lam et al. compared the retinal nerve fiber layer measurements of attack eyes and their fellow eyes after a single unilateral attack of acute primary angle closure (APAC) using scanning laser polarimetry six months after the acute attack8. Retinal nerve fiber layer damage was documented in eyes where the duration of the APAC attack lasted more than 48 hours8. Decompression retinopathy following laser peripheral iridoplasty for acute primary angle closure was reported in two cases reported by Lai, Lee, Leung and Chung.9 In order to compare the efficiency of laser peripheral iridoplasty and medical treatment, as well as to identify any morbidity that may come from sudden decompression of the eye, we undertake this randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 21 years with ability to give informed consent and cooperate for a slit lamp laser procedure
* Subjects at their first presentation of acute primary angle closure attack.
* Intraocular pressure levels of 40 mm Hg or higher by applanation tonometry or tonopen
* Pupillary block as the main mechanism of angle closure
* No previous treatment

Exclusion Criteria:

* Age less than 21 years
* Angle closure due to non-pupil block mechanism (e.g. plateau iris, pseudoplateau, phacomorphic, malignant glaucoma) or other secondary causes (subluxed lens, neovascular, uveitic, traumatic, post-operative)
* Angle closure patients whose IOP's are not lowered by 20% or more, and are unresponsive to maximum medical IOP-lowering agents after one hour of initiating treatment and needing other intervention/s to lower IOP(e.g. iridoplasty, surgery).
* Corneal opacities or abnormalities obstructing laser application
* Use of contact lens
* Single-eyed patients

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-02; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
optic nerve head stereometric analysis HRT3 and Stratus OCT,optic nerve head and RNFL & macula thickness average. AGIS scores of HVF is the measure of functional status. | 1 year

SECONDARY OUTCOMES:
amount and rate of IOP-lowering,gonioscopy and ASOCT changes, change in LOCS grading for cataract, corneal decompensation & edema,macular,retinal edema by Stratus OCT. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul TK Chew, A/Prof, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, 5 Lower Kent Ridge Road, Singapore, Singapore

REFERENCES:
- [Background] Lai JS, Tham CC, Chua JK, Poon AS, Lam DS. Laser peripheral iridoplasty as initial treatment of acute attack of primary angle-closure: a long-term follow-up study. J Glaucoma. 2002 Dec;11(6):484-7. doi: 10.1097/00061198-200212000-00005. PMID 12483091